CLINICAL TRIAL: NCT02473679
Title: Influence of the Education in Layperson Resuscitation and Preparation the Patrol Car of the City Police With Automatic External Defibrillators and Automated Ventilation Equipment on Out of Hospital Resuscitation Outcome
Brief Title: Influence of the Education in Layperson in Out of Hospital Resuscitation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK2014 - 0665
Record Dates: First submitted 2015-05-13; First posted 2015-06-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Arrest, Sudden; Heart Arrest
Keywords: First Responder; BLS; AED; Resuscitation
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac arrest occurs frequently and the outcome after out-of-hospital resuscitation is often fatal. Disturbing is that more than half of the surviving patients suffer from permanent impairment of cognitive functions, such attention, memory and executive functioning. With all the efforts to achieve a high quality initial resuscitation management the time delay between cardiac arrest and the beginning the initial resuscitation maneuver is the main reason for the still poor outcome. To shorten this fatal time delay, current efforts of national and supranational health authorities aime at the non-medically trained lay person, who should carry out basic life support directly on the scene supported by the use of public available semi-automatic defibrillators (AED).

DETAILED DESCRIPTION:
It is a combined retrospective and prospective observational single center study. Data of all Out of Hospital patients suffered a cardiac arrest in Zurich city will be collected according to the Utstein criteria. The aim of this study is to investigate the impact of trained police forces in the resuscitation outcome.

ELIGIBILITY:
Inclusion Criteria:

* All Out of hospital patients suffering cardiac arrest in Zurich City, resuscitated by lay persons, city police and or trained emergency medical services

Exclusion Criteria:

* individuals with cardiac arrest occurring in the presence of EMS
* individuals in whom there were apparent toxic, traumatic or suicidal etiologies for unconsciousness
* drowned individuals and individuals with terminal illness
* documented negation of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out of hospital patients suffered or suffering cardiac arrest, who were or will be resuscitated by laypersons, city police and/or trained emergency medical services teams who were called to the emergency
Sampling Method: Probability Sample
Enrollment: 1662 (Actual)
Dates: Start 2003-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time line for restoration the circulation | participants will be followed from origin of the event up to 12 month or death
  Timeline for restoration the circulation after layperson started the reanimation

SECONDARY OUTCOMES:
Time interval to first shock , | participants will be followed from origin of the event up to 12 month or death
  Time interval from the emergency call to first shock for ventricular fibrillation
Neurologic outcome | participants will be followed from origin of the event for duration of hospital stay, follow up after 12 month or death
  Data will be collected according to Utstein criteria
Time interval removal from ICU as well as discharged from hospital | participants will be followed from origin of the event up to 12 month or death
  Time interval up to the removal from ICU as well as duration of hospital stay
Definitive survival rate | participants will be followed from origin of the event up to 12 month or death
  Survival rate of participants resuscitated by layperson after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Donat R Spahn, Prof, Principal Investigator — IFA, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland